CLINICAL TRIAL: NCT06861777
Title: Clinical Trial of Total Neoadjuvant Therapy Combined With Adebrelimab in Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Total Neoadjuvant Therapy Combined With Adebrelimab in Locally Advanced Resectable ESCC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: YIN LI (Other)
Responsible Party: Sponsor-Investigator, YIN LI, Head of the Department of Esophageal and Mediastinal Surgery at Cancer Hospital, Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5115
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: locally advanced resectable ESCC; adebrelimab; total neoadjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Clinical Trials, Phase II as Topic; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TNT group one (phase 2) (Experimental): Neoadjuvant adebrelimab combined with paclitaxel/nab-paclitaxel and cisplatin for 2 cycles, followed by chemoradiotherapy (paclitaxel/nab-paclitaxel and cisplatin+41.4Gy/23f), and then surgical resection 4-8 weeks later.
  Interventions: Other: Adebrelimab + paclitaxel/nab-paclitaxel + cisplatin followed by chemoradiotherapy
- TNT group two (phase 2) (Experimental): Neoadjuvant chemoradiotherapy (paclitaxel/nab-paclitaxel and cisplatin+41.4Gy/23f), followed by adebrelimab combined with paclitaxel/nab-paclitaxel and cisplatin for 2 cycles, and then surgical resection 4-8 weeks later.
  Interventions: Other: chemoradiotherapy followed by adebrelimab + paclitaxel/nab-paclitaxel + cisplatin
- TNT treatment group (phase 3) (Experimental): The patients received neoadjuvant TNT treatment, followed by surgical resection 4-8 weeks later, and then adjuvant adebrelimab for one year.
  Interventions: Other: TNT treatment [TNT group one (phase 2) or TNT group two (phase 2)]
- CRT treatment group (phase 3) (Active Comparator): Neoadjuvant chemoradiotherapy (paclitaxel/nab-paclitaxel and cisplatin+41.4 Gy/23f), followed by surgical resection 4-8 weeks later. Non-pCR subjects received adjuvant treatment with adebrelimab for one year.
  Interventions: Other: Chemoradiotherapy

INTERVENTIONS:
Other: Adebrelimab + paclitaxel/nab-paclitaxel + cisplatin followed by chemoradiotherapy — Neoadjuvant treatment:
  adebrelimab 1200 mg/m2 d1+ paclitaxel d1/nab-paclitaxel d1,8, + cisplatin d1, Q2W×2 followed by chemoradiotherapy (paclitaxel /nab-paclitaxel + cisplatin + 41.4Gy/23f), surgical resection 4-8 weeks later neoadjuvant treatment.
  Arms: TNT group one (phase 2)
Other: chemoradiotherapy followed by adebrelimab + paclitaxel/nab-paclitaxel + cisplatin — Neoadjuvant treatment:
  chemoradiotherapy (paclitaxel /nab-paclitaxel + cisplatin + 41.4Gy/23f), followed by adebrelimab 1200 mg/m2 d1+ paclitaxel d1/nab-paclitaxel d1,8, + cisplatin d1, Q2W×2 surgical resection 4-8 weeks later neoadjuvant treatment.
  Arms: TNT group two (phase 2)
Other: TNT treatment [TNT group one (phase 2) or TNT group two (phase 2)] — Neoadjuvant treatment:
  TNT treatment [TNT group one (phase 2) or TNT group two (phase 2)] followed by surgical resection 4-8 weeks later adjuvant treatment: adebrelimab 1200 mg/m2 d1, W3Q, adjuvant treatment for one year
  Arms: TNT treatment group (phase 3)
Other: Chemoradiotherapy — Neoadjuvant treatment:
  chemoradiotherapy (paclitaxel 50 mg/m2/nab-paclitaxel 60 mg/m2 d1, 8, 15, 22,29 + cisplatin 25 mg/m2 d1, 8, 15, 22,29 + 41.4Gy/23f), followed by surgical resection 4-8 weeks later. adjuvant treatment: non-pCR: adebrelimab 1200 mg/m2 d1, W3Q, adjuvant treatment for one year pCR: observation
  Arms: CRT treatment group (phase 3)

SUMMARY:
Esophageal cancer is a malignant tumor with high incidence rate and mortality in China. According to the data of the World Health Organization, 324000 new cases and 301000 deaths of esophageal cancer will occur in China in 2020, accounting for 53.70% and 55.35% of the global incidence and death of esophageal cancer respectively.

Surgery is the main method for locally advanced resectable esophageal cancer, combined with chemoradiotherapy(CRT), in order to achieve curative resection. However, after neoadjuvant chemoradiotherapy and surgery, 36-50% of patients still experience recurrence or metastasis, and the prognosis for early recurrence is worse. Adjuvant chemotherapy plays a particularly beneficial role in terms of disease-free survival(DFS) in patients who did not receive neoadjuvant therapy and patients with pathologic lymph-node-positive disease. however, less than 50% of eligible patients receive their scheduled adjuvant chemotherapy due to delays, treatment compliance, and postoperative complications. Among patients with resected esophageal cancer who had received neoadjuvant CRT, DFS was significantly longer among those who received nivolumab adjuvant therapy than among those who received placebo.

Total neoadjuvant therapy (TNT), attempts to deliver both systemic chemotherapy and neoadjuvant CRT prior to surgery, which may become a new treatment direction for patients with locally advanced resectable esophageal cancer. Ongoing progress in all treatment modalities involved in TNT holds the promise to enhance further the outcomes of patients with esophageal cancer. Immunotherapy, as a breakthrough therapy in the systemic treatment of advanced esophageal cancer, has become an indispensable component of the exploration of TNT model. Currently, several prospective exploratory studies suggest that immunotherapy combined with TNT can improve the pCR rate of esophageal cancer patients, achieving good short-term efficacy and tolerable safety.

However, further exploration is needed for the combination of immunotherapy and TNT. This study first explores the efficacy and safety of two types of total neoadjuvant therapy in phase II: the combination of adebrelimab and chemotherapy followed by chemoradiotherapy, or the combination of adebrelimab and chemotherapy after chemoradiotherapy. A more promising treatment plan will be selected for a phase III randomized controlled trial and confirm the superiority of adebrelimab combined with TNT over neoadjuvant CRT in terms of pathological complete response overall survival in patients with locally advanced resectable esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a informed consent form and voluntarily join this study;
2. Esophageal squamous cell carcinoma diagnosed by histopathology or cytology;
3. Diagnosed as thoracic esophageal cancer by CT/MRI/EUS and clinically staged as T1b-3N1-2M0 or T3N0M0 (according to AJCC 8th edition);
4. Expected to achieve R0 resection;
5. Age ≥ 18 years old, regardless of gender;
6. ECOG PS 0-1;
7. Have not received any anti-tumor treatment for esophageal cancer in the past;
8. Plan to undergo surgical treatment after completion of neoadjuvant therapy;
9. No surgical contraindications;
10. The main organ functions are normal, including:

    1. Blood routine examination:

       neutrocyte count ≥ 1.5 × 109/L Platelet count ≥ 100 × 109/L Hemoglobin ≥ 90 g/L
    2. Blood biochemistry test:

       Total bilirubin ≤ 1.5 × ULN ALT ≤ 2.5×ULN，AST ≤ 2.5×ULN， Serum creatinine ≤ 1.5 × ULN, or creatinine clearance rate ≥ 50 mL/min (Cocheroft Gault formula, see Appendix 2)
    3. Coagulation function:

    INR ≤ 1.5 × ULN APTT ≤ 1.5 × ULN
11. Women who have the ability to conceive or men whose spouses have the ability to conceive should use effective contraceptive measures during the study period;
12. The subjects showed good compliance and cooperated with follow-up visits;

Exclusion Criteria:

1. Tumors or lymph nodes significantly invade adjacent organs of esophageal lesions;
2. Patients with supraclavicular lymph node metastasis;
3. Individuals at risk of perforation, fistula, etc;
4. There are uncontrollable pleural effusion, pericardial effusion, or ascites that require repeated drainage;
5. Poor nutritional status, BMI < 18.5 Kg/m2；
6. Have a history of allergies to monoclonal antibodies, any components of Adebrelimab, paclitaxel, cisplatin, or other platinum based drugs in the past;
7. Have received or are currently receiving any of the following treatments:

   1. Any radiotherapy, chemotherapy, or other anti-tumor drugs targeting tumors;
   2. Within 2 weeks prior to the first use of the investigational drug, immunosuppressive or systemic hormone therapy was being used to achieve immunosuppressive effects;
   3. Received attenuated live vaccine within 4 weeks prior to the first use of the investigational drug;
   4. Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
8. Suffering from any active autoimmune disease or history of autoimmune disease;
9. History of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation;
10. There are clinical symptoms or diseases of the heart that have not been well controlled;
11. Severe infection (CTCAE>grade 2) occurred within 4 weeks prior to the first use of the investigational drug;
12. Discovery of active pulmonary tuberculosis infection through medical history or CT examination;
13. Active hepatitis B and hepatitis C exist;
14. Diagnosed with other malignant tumors within 5 years prior to the first use of the investigational drug;
15. Pregnant or lactating women;
16. According to the researchers' assessment, there are other factors that may lead to the forced termination of the study midway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
pCR (phase 2 and phase 3) | one month after esophageal cancer surgery
  The rate of patients with primary tumor and lymph nodes both achieved pathological complete response
EFS (phase 3) | Approximately 5 years
  The time from randomization to the occurrence of events as defined by the study protocol.

SECONDARY OUTCOMES:
R0 resection rate (phase 2 and phase 3) | one month after esophageal cancer surgery
  The proportion of patients with negative surgical margins among those who underwent radical surgery for esophageal cancer.
MPR (phase 2 and phase 3) | one month after esophageal cancer surgery
  The percentage of subjects with less than 10% tumor residue in the primary tumor site.
Tumor regression (phase 2 and phase 3) | one month after esophageal cancer surgery
  The research center performed tumor regression grade (TRG) assessments using the Mandard 5-point classification system.
ypTNM (phase 2 and phase 3) | one month after esophageal cancer surgery
  According to AJCC 8th Edition criteria, the rate of patients who have reached ypI-IVA stages respectively.
OS (phase 2 and phase 3) | Approximately 6 years
  The time from randomization to death due to any cause.
EFS (phase 2) | Approximately 5 years
  The time from randomization to the occurrence of events as defined by the study protocol.
DFS (phase 3) | Approximately 5 years
  For postoperative subjects free of esophageal cancer disease, the time from the first day without disease (i.e., the date of surgery) to either local recurrence or distant metastasis, or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After the conclusion of the study, Individual Participant Data (IPD) will be shared through the publication of articles.
Supporting Information: Study Protocol, SAP
Time Frame: After the study concludes, please contact the principal investigator for specifics.
Access Criteria: Please contact the principal investigator.